CLINICAL TRIAL: NCT03046030
Title: Mechanistic Studies on Video-guided Acupuncture Imagery Treatment of Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jian Kong, Associate Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016P001293
Record Dates: First submitted 2017-01-27; First posted 2017-02-08 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy Volunteers (Experimental): In this experiment, we will apply a crossover design in healthy subjects. Each subject will receive four treatments in four separate sessions: 1) VGAIT, 2) VGAIT control condition, 3) real acupuncture, and 4) sham acupuncture. Each session will be separated by at least 7 days. Subjects will participate in five experimental sessions: a training and familiarity behavioral session and four fMRI sessions during which the subject will receive one of the four treatments.
  Interventions: Other: Real acupuncture; Other: Sham acupuncture; Other: VGAIT; Other: VGAIT control

INTERVENTIONS:
Other: Real acupuncture — Verum acupuncture will be applied on the right SP6 and SP9. For each subject, leg position, acupoint location, and needling parameters (1-2 cm depth, 120 rotations / minute, 90˚ insertion angle, moderate deqi sensations on a 0-10 scale) will be kept constant. For the low dose acupuncture group, needles will be rotated at one point and then the other in 15-second rotations with 20-30 second breaks. The specific starting acupoint will be randomized across subjects but kept consistent for each subject across sessions.
Other: Sham acupuncture — Placebo acupuncture will be applied at two sham points using specially designed sham acupuncture needles [20, 35, 104-106]. The sham needles differ from regular needles by possessing blunt and retractable tips. Instead of penetrating the skin, the point of the Streitberger needle retracts up the handle shaft when the acupuncturist presses it against the skin. This sham device has been validated by studies showing that subjects cannot distinguish between genuine and sham needling [20, 35, 104]. Two sham points will be used during placebo acupuncture: sham point 1 is located 1 cun posterior to the superior 1/3 of K9 and K10. Sham 2 is located 1 cun posterior to K8. Both points are located on the leg where there is no meridian passing through. Sham acupuncture treatment will be the same as verum acupuncture.
Other: VGAIT — In Session 1, all patients will first be introduced to acupuncture treatment, particularly the sensation evoked by acupuncture needles. This will be followed by a five-minute acupuncture exposure applied by a licensed acupuncturist. The exposure will include multiple acupuncture needle manipulations across the two acupoints (SP 6 and SP 9) used in this study. The paradigm applied will be identical to real acupuncture treatment, and the procedure will also be video recorded for the following session. At the beginning of the VGAIT session, patients will be trained for imagery acupuncture outside the fMRI scan. Subjects will first read a script introducing the imagery acupuncture treatment. Then, VGAIT will be applied during scanning. Identical to the acupuncture treatment, there are two fMRI scans during VGAIT, each lasting about 10 minutes. We will ask the patient to measure the sensations they feel during treatment using the MGH Acupuncture Sensation Scale (MASS) after treatment.
Other: VGAIT control — The control condition will be the same as VGAIT, except we will use cotton swabs repeatedly touching at non-acupoints with a frequency of about 1 Hz using the same paradigm of verum / sham acupuncture. They will also read a script describing what they are about to see. Then, VGAIT control will be applied during scanning. We will ask the patient to measure the sensations they feel during treatment using the MASS after treatment.

SUMMARY:
The aim of this proposal is to investigate brain response and connectivity changes evoked by video-guided acupuncture imagery treatment (VGAIT) and verum and sham acupuncture in healthy and patient populations to elucidate the underlying brain mechanisms of mind-body interaction, imagery, and acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* Right handed healthy male and female adults aged 18-60
* No contraindications to fMRI scanning

Exclusion Criteria:

* Current or past history of major medical, neurological, or psychiatric illness
* Any pain disorder
* Pregnancy
* Non-fluent speaker of English

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
fMRI signal increases | 4 days; Sessions 2-5

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No